CLINICAL TRIAL: NCT05282186
Title: What the Nose Knows: Hedonic Capacity, Psychosocial Interventions and Outcomes in Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Raquelle Mesholam-Gately, Assistant Professor of Psychology, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022P000199; R21MH127479-01A1 (NIH)
Record Dates: First submitted 2022-03-02; First posted 2022-03-16 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Schizophrenia
Keywords: olfaction; reward
MeSH Terms: conditions — Schizophrenia; Anosmia

STUDY DESIGN:
Intervention Model Description: Randomized cluster design with 19 service centers assigned to one of the two treatments.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cognitive Enhancement Therapy (Experimental): CET is a comprehensive manualized cognitive remediation program designed to maximize gains in social functioning by integrating computer-based training to enhance neurocognition with group-based exercises to improve social cognition.
  Interventions: Behavioral: Cognitive Enhancement Therapy
- Social Skills Training (Active Comparator): The HOPES social rehabilitation program uses the principles of SST (modeling, role playing, positive and corrective feedback, homework assignments, in vivo skills practice), designed to improve both psychosocial functioning and preventive health.
  Interventions: Behavioral: Social Skills Training

INTERVENTIONS:
Behavioral: Cognitive Enhancement Therapy — CET's group-based exercises are delivered for 1.5 hours each week in a group of 6-8 participants led by a clinician and an assistant, for one year. During each of three modules (basic concepts, social cognition, CET applications), the groups focus on acquisition of adult social milestones in perspective-taking, social context appraisal, and other aspects of social cognition, with psychoeducational lectures, homework assignments, and in-group exercises. Weekly supervision sessions for the clinician trainers will include review of how patients respond to the different demands of computer-based training and group-based exercises and guidance about improving engagement in both.
  Arms: Cognitive Enhancement Therapy
Behavioral: Social Skills Training — The psychosocial component involves weekly skills training classes delivered over one year, with modules including "Communicating Effectively," "Making and Keeping Friends," "Making the Most of Leisure Time," "Healthy Living," "Using Medications Effectively," and "Making the Most of a Health Care Visit" (Pratt et al., 2008). Participants attend two sessions each week (normally morning and afternoon of the same day): a 90-minute session focused on a specific skill and a 60-minute session in which the specific skill is used in role-play exercises.
  Other Names: HOPES
  Arms: Social Skills Training

SUMMARY:
This project proposes to conduct the first study of the predictive utility of olfactory hedonic measurement for targeted psychosocial rehabilitation in schizophrenia. The information gathered from the project is of considerable public health relevance, in that, through simple, reliable olfactory assessment, it will provide knowledge about which individuals are most likely to benefit from these psychosocial interventions. Such information is crucial for tailoring existing interventions and developing new approaches to optimize outcomes in schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

1. age 18 to 65;
2. DSM-5 diagnosis of schizophrenia or schizoaffective or schizophreniform disorder

Exclusion Criteria:

1. the presence of a current organic brain syndrome;
2. a current and severe substance use disorder (DSM-5);
3. intellectual disability (DSM-5)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2022-09-02 (Actual); Primary Completion 2025-05-31 (Actual); Study Completion 2025-05-31 (Actual)

PRIMARY OUTCOMES:
Change in Social Adjustment Scale II | Measurement at 0, 6, 12 months
  Measure of ability to engage socially in community settings
Change in Heinrich Quality of Life Scale | Measurement at 0, 6, 12 months
  Measure of quality of life
Change in Social Skills Performance Assessment rating scale | Measurement at 0, 6, 12 months
  Social skills measure using role plays

SECONDARY OUTCOMES:
Change in NIH Toolbox® for Assessment of Neurological and Behavioral Function (NIH Toolbox) | Measurement at 0, 6, 12 months
  Neurocognition
Change in Managing Emotions subscale of the Meyer-Salovey-Caruso Emotional Intelligence Test (MSCEIT) | Measurement at 0, 6, 12 months
  Social cognition

CONTACTS AND LOCATIONS:
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No